CLINICAL TRIAL: NCT00780117
Title: Characterization of At-risk Population and Prognosis Factors for SACRO-coccygeal Teratoma in CURRARINO Syndrome. A Clinical, Molecular and Pathological Study.
Brief Title: Characterization of At-risk Population for Pre-sacral Tumor in CURRARINO Syndrome
Acronym: Currarino
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P070305
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: CURRARINO Syndrome; Sacrococcygeal Teratoma; Presacral Mass
Keywords: CURRARINO syndrome; Sacrococcygeal teratoma; HLXB9 (MNX1) gene; Alpha foeto protein; Prognosis factors
MeSH Terms: conditions — Currarino triad

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pathological tumoral tissue analysis after surgical removal · Annual serum alpha-foeto protein level monitoring
Oversight: Data Monitoring Committee: No

SUMMARY:
Contribute to support hypothesis of relationships between genes involve in oncogenesis and those involve in embryological development.

DETAILED DESCRIPTION:
CURRARINO syndrome (CS) (OMIM 176450) is a rare congenital disease described in 1981, as the association of, at least, three main clinical features: typical sacral malformation (sickled-shape sacrum or total sacral agenesis below S2), hindgut anomalies and pre-sacral tumor. To date, neurological defects, as tethered cord and/or lipoma of the filum or the conus, are up lighted to be as a fourth major clinical sign.In half of cases, CS is ascribed to heterozygous mutations of the HLXB9 gene (or MNX1 gene, OMIM 142994) located at 7q36, with an autosomal dominant mode of inheritance. The HLXB9 gene is involved in motoneurons and caudal development of the embryo. However, genetic heterogeneity is suspected, since patients without HLXB9 mutation harbour subtle phenotypic variations. Presently, no other locus has been identified. The pre-sacral tumor develops in almost 80% of CS. When it is a teratoma (30% of cases), it may turn into malignancy in 1 to 4 % of cases, according to literature. As far as we know, no clinical, molecular or pathological marker is operational to predict tumoral evolution and give any prognosis. Major aim of this study is to find out any correlation between clinical signs, constitutional and somatic genetic anomalies of HLXB9 gene and other candidate genes, and/or pathological features and tumoral evolution in CS. Evaluation of the pre-sacral tumor evolution is based on local recurrence or distance metastasis after surgical removal. Annual serum alpha-foeto-protein level monitoring is also performed, as the unique marker of teratoma.This study specifically required annual clinical examination and lumbar-sacral MRI imaging, three blood samples at inclusion and an annual blood sample.This multicentric study will last for at least 6 years. Eighty patients will be included and follow up for at least 3 years. Finally, this study may help identify a group of at-risk patients for tumor development and malignant transformation if pre-sacral teratoma. It will also help define objective clinical, radiological, molecular, pathological and/or biological criteria for long lasting survey. In general, it may also contribute to support hypothesis of close relationships between genes involve in oncogenesis and those involve in embryological development.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 out of the 4 major signs of CURRARINO syndrome:

  1. Sacral agenesis
  2. Hindgut malformation or chronic constipation
  3. Presacral tumor and/or
  4. TETHECORD syndrome and/or lipoma of the filum or the conus
* Anomaly genotyping HLXB9 without clinical expression

Exclusion Criteria:

- Opposition to sign informed consent agreement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: specialized consultations in the currarino syndrom network
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Annual lumbar-sacral MRI is performed | one year

SECONDARY OUTCOMES:
Pathological tumoral tissue analysis after surgical removal | 3 years
Annual serum alpha-foeto protein level monitoring | one year

CONTACTS AND LOCATIONS:
Overall Officials: Celia CRETOLLE, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades Pediatric Surgery Department, Paris, France